CLINICAL TRIAL: NCT00000984
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant CD4 (rCD4) in Infants and Children Infected With or at Risk for HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 101; CO102G
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Acquired Immunodeficiency Syndrome; Antigens, CD4; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — CD4 Antigens

INTERVENTIONS:
Drug: CD4 Antigens

SUMMARY:
AMENDED: As of 10/19/90 only Children 0 to 3 months are being enrolled. Original design: To determine whether the experimental drug recombinant CD4 (rCD4), which is produced through genetic engineering technology, is safe and well-tolerated in children infected with or at risk for HIV infection.

rCD4 may be an effective treatment for HIV infection, based on its ability to block infection of human cells by HIV in laboratory tests. However, the activity of rCD4 still needs to be confirmed in clinical trials. It is hoped that these tests will show that rCD4 is both safe and effective in treating children who are infected with or who are at risk for infection with HIV.

DETAILED DESCRIPTION:
rCD4 may be an effective treatment for HIV infection, based on its ability to block infection of human cells by HIV in laboratory tests. However, the activity of rCD4 still needs to be confirmed in clinical trials. It is hoped that these tests will show that rCD4 is both safe and effective in treating children who are infected with or who are at risk for infection with HIV.

Children have preliminary testing and evaluation to determine eligibility and health. The dosage schedule varies with the dose. During the course of the study, children are monitored for safety through physical exams and blood tests. They have blood withdrawn to study the response to rCD4 and measure the activity of rCD4 in the body. Children may receive immunization of DPT (diphtheria, pertussis, tetanus) or DT and a polio vaccine to measure their antibody response. If the rCD4 is beneficial, children may continue treatment. The study is conducted in four parts:

* Part A: Children 13 to 18 years old.
* Part B: Children 3 months to less than 13 years old.
* Part C: Full-term infants over 3 months old.
* Part D: Preterm infants less than 3 months old. Parts C and D are not started until parts A and B have been completed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic medication for patients with previous documented episodes of Pneumocystis carinii pneumonia (PCP).
* Concomitant zidovudine (AZT) or intravenous gamma globulin (IVIG) during maintenance therapy phase of the study.

AMENDED: As of 10/19/90 only Children 0 to 3 months are being enrolled.

Original design: Patients must be infected with HIV or at risk for HIV infection. They must be one of the following:

* Asymptomatic.
* Mildly symptomatic but not eligible for and/or decline ACTG protocol 052.
* Markedly symptomatic but not eligible for and/or decline ACTG protocol 051 or cannot tolerate zidovudine (AZT) therapy.

All patients must have:

* A life expectancy of at least 3 months.
* A legally-qualified guardian with the ability to sign a written informed consent form, which must be obtained prior to treatment. A willingness to abstain from all other experimental therapy for HIV infection during the entire study period.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Intravenous gamma globulin (IVIG).
* Pentamidine.
* Trimethoprim / sulfamethoxazole (TMP/SMX).
* Corticosteroids.
* Nonsteroidal anti-inflammatory agents (NSAIDS).
* Other known immunomodulatory agents.
* All other experimental therapies.

Patients will be excluded from the study for the following reasons:

* Serious active opportunistic infection or malignancies prior to study entry.
* Defined organ insufficiencies.

Prior Medication:

Excluded within 3 weeks of study entry:

* Zidovudine (AZT).
* Intravenous gamma globulin.
* Cancer chemotherapy.
* Immunomodulatory agents.
* Other experimental therapy.

Patients may not have any of the following diseases or symptoms:

* Serious active opportunistic infection or malignancies prior to study entry.
* Cardiopathy.
* Two or more episodes of prior Pneumocystis carinii pneumonia (PCP).
* Hematologic insufficiency defined as granulocytes = or < 1000 cells/mm3; platelets = or < 100000 cells/mm3; hemoglobin = or < 8 g/dl.
* Renal insufficiency defined as creatinine > 2 mg/dl; = or > 5 white blood cells or red blood cells/hpf or = or > 2+ proteinuria in urine.
* Hepatic insufficiency defined as bilirubin = or > 3 x upper limit of normal; SGOT = or > 10 upper limit of normal.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: P Weintrub, Study Chair
Locations (6):
- United States (6):
  - Northern California Pediatric AIDS Treatment Ctr / UCSF, San Francisco, California
  - Stanford Univ School of Medicine / Pediatrics, Stanford, California
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Children's Memorial Med Ctr, Chicago, Illinois
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Weintrub P, Yogev R, Conner E, Wilfert K, Mordenti J, Ammann AJ. Safety and pharmacokinetics of recombinant CD4 in children with HIV infection. Int Conf AIDS. 1990 Jun 20-23;6(2):95 (abstract no FB23)